CLINICAL TRIAL: NCT05450081
Title: Clinical Trials to Evaluate the Association Between the Results of Specific Genetic Tests and the Efficacy of Targeted Therapies in Patients With Non-small Cell Lung Cancer
Brief Title: Association Between the Results of Specific Genetic Tests and the Efficacy of Targeted Therapies in Patients
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Other Study IDs: ART
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aimed to evaluate the correlation between test reagent specific gene test results and the efficacy of relevant targeted drugs in patients with non-small cell lung cancer, and to support the continued registration of test reagents.

ELIGIBILITY:
Inclusion Criteria:

* 1)≥18，advanced non-small cell lung cancer confirmed by histopathology, and were previously or currently treated with gefitinib tablets (as the first-line treatment) or osimertinib (first-generation TKI resistance treatment) or crizotinib capsules monotherapy were evaluated for efficacy.
* 2) Able to provide FFPE samples with a storage life of 5 years: Large specimen 5 pieces in each case; 10 puncture specimens in each case

Exclusion Criteria:

* 1) Pathological evaluation of the tissue sample has too few tumor cells (total number of tumor cells >20%);
* 2) Combination therapy with chemotherapy/radiotherapy/other targeted drugs/immunotherapy drugs;
* 3) Maintenance treatment when the disease does not progress after other anti-tumor treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer who have previously received single-agent K therapy
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
PFS | October 2022-December 2022
  Progression free survival time
ORR | October 2022-December 2022
  Objective response rate
Consistency | October 2022-December 2022
  he consistency of efficacy between specified kit and 22C3

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China